CLINICAL TRIAL: NCT03397537
Title: Letrozole as Neoadjuvant Treatment in Postmenopausal and Premenopausal Patients With Highly Endocrine Responsive Operable Breast Cancer
Brief Title: Neoadjuvant Endocrine Therapy in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170811
Record Dates: First submitted 2017-12-25; First posted 2018-01-12 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2012-09

CONDITIONS: Highly Endocrine Responsive Operable Breast Cancer
Keywords: Breast Neoplasms Endocrine-responsive Neoadjuvant Duration Letrozole
MeSH Terms: interventions — Letrozole; Tablets; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the postmenopausal (Other): 2.5 mg letrozole every day for six months
  Interventions: Drug: Letrozole 2.5Mg Tablet
- the premenopausal (Experimental): 2.5 mg letrozole daily along with a GnRH analogue for ovarian suppression, which was administered as an intramuscular injection of 3.75 mg triptorelin every 28 days for 6 months.
  Interventions: Drug: Letrozole 2.5Mg Tablet; Drug: GnRH analogue

INTERVENTIONS:
Drug: Letrozole 2.5Mg Tablet — letrozole 2.5mg p.o.qd
Drug: GnRH analogue — 3.75 mg triptorelin im. q28d
  Arms: the premenopausal

SUMMARY:
The study aimed to compare the duration to complete or partial response (CR/PR) and the overall response rates (ORR) after six months of neoadjuvant endocrine therapy between pre-menopausal group and post-menopausal group with highly endocrine responsive operable mammary carcinoma.

DETAILED DESCRIPTION:
Estrogen receptor (ER) positive constitutes about 75% of all breast cancer(BC). Neoadjuvant endocrine therapy(NET) plays an important part in primary therapy of the hormone receptor (HR) -positive and HER2 -negative breast cancer. Recent studies revealed that the third-generation aromatase inhibitors (AIs) have superior ORR than tamoxifen in the HR-positive BC post-menopausal patients. The Z1031 trial showed that Letrozole obtained better ORR than the other two AIs anastrozole and exemestane after 16-18 weeks NET, although without any statistically significance.

In spite of these findings, the optimal duration of NET has not been fully elaborated, Although prolonged treatment might further reduce the tumor size. Further clinical benefits were achieved when the period of treatment of neoadjuvant letrozole prolonged more than three to four months. The 2015 St. Gallen International Consensus Conference recommended continuing neoadjuvant therapy in highly hormone-sensitive breast cancer for a minimum of 4-8 months. However, most studies aim to identify the excellent efficacy of the AIs compared with other drugs but not the duration of NET therapy. Antonio et al. suggest that the time to maximum clinical efficacy may be the optimal period of treatment for the patients; And the median time to maximum efficacy was 4.2 months (95% CI, 4.0-4.5). The present study evaluated the time to CR/PR and the ORR after 6 months of NET.

Previous clinical studies investigating NET mainly focused on post-menopausal women, data on pre-menopausal women is still relatively lacking due to the widely perception that more benefit may be achieved from neoadjuvant chemotherapy (NCT) among younger patients. The result of Z1031 trial showed superiority of neoadjuvant of AIs and promoted wider application of AIs as NET in the HR-positive post-menopausal women, and the clinical response rate (CRR) of letrozole was 74.8% after 16-18 weeks of treatment. The combination of AIs and GnRH analogue may be alternative for selected pre-menopausal patients. The STAGE trial showed the overall response rates of anastrozole plus goserelin in pre-menopausal patients was 70.4% after 6 months of NET. However, studies comparing the ORR and optimal duration of NET between pre-menopausal and post-menopausal patients were rare.

The purpose of the our research was to compare the duration to CR/PR and the ORR after 6 months of NET between pre-menopausal and post-menopausal women with highly endocrine responsive operable BC.

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥18 years
2. ER-positive (≥50%), PgR-positive (≥50% ), HER2-negative, and previously untreated, non-metastatic primary invasive BC.
3. The tumour size had to be >1 cm.

Exclusion Criteria:

1. male patients;
2. patients with inflammatory breast cancer or distant metastasis;
3. patients who were previously treatment treated with chemotherapy, radiation therapy or prior treatment with AIs or antiestrogens for breast cancer;
4. patients with a second concomitant neoplasm;
5. patients who could not meet the eligibility criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
ORR | six months
  overall response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Minyi Cheng, Guanzhou, Guangdong, China